CLINICAL TRIAL: NCT04428450
Title: Internet-Based Treatment of Depression: A Randomized Controlled Trial Comparing Guided With Unguided Self-Help
Brief Title: Internet-Based Treatment of Depression: Comparing Guided With Unguided Self-Help
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia AG (Industry)
Collaborators: University of Bern (Other); Linkoeping University (Other Government); Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Berger_2011_deprexis
Record Dates: First submitted 2020-06-09; First posted 2020-06-11 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Deprexis (unguided) (Experimental): web-based self-help program without any support from a therapist during the 10-week treatment period
  Interventions: Device: Deprexis
- Deprexis (guided, with therapist) (Experimental): web-based self-help program plus scheduled e-mail contact with a therapist during the 10-week treatment period
  Interventions: Device: Deprexis
- Wait-list (No Intervention): Wait-list group (subjects receive access to Deprexis after 10 weeks)

INTERVENTIONS:
Device: Deprexis — CBT-based, integrative online self-help program
  Arms: Deprexis (guided, with therapist); Deprexis (unguided)

SUMMARY:
The study is a randomized controlled trial and to compare the benefits of a 10-week web-based unguided self-help treatment with the same intervention complemented with weekly therapist support via e-mail. A waiting-list control group will be included. The Beck Depression Inventory (BDI-II) will be used as the primary outcome measure. Secondary outcomes include general psychopathology, interpersonal problems, and quality of life.

DETAILED DESCRIPTION:
Depression is a major health problem associated with significant disability and economic costs. Although depression can be treated effectively with several psychological and pharmacological treatment options, many sufferers still seek or receive inadequate therapy or no therapy at all. Internet-based treatments may help to serve this demand, being accessible anytime and anywhere making it easier for underserved populations and people living in remote areas to receive treatment. The present study aims to assess the efficacy of an internet-based CBT intervention for depression (Deprexis), directly comparing the benefits of a low intensity therapist-guided with an unguided self-help version. A waiting-list control group will be included. Individuals meeting the diagnostic criteria of major depression or dysthymia will be randomly assigned to one of the three conditions. While unguided self-help will not include any contact with a therapist or the study team during the treatment, guided self-help will include a weekly scheduled e-mail feedback by a therapist and the possibility to ask questions via e-mail. While in an earlier study Deprexis was assessed as an add-on to TAU, this study will examine the efficacy of the program when delivered as a stand-alone intervention (i.e., only individuals who currently do not receive psychotherapy will be included). Moreover, this study will include a structured diagnostic interview at pretreatment. Only participants fulfilling the criteria of a depressive disorder (major depression or dysthymia) will be included in the trial. Participants will be recruited in Switzerland and Germany via articles in national and regional newspapers and a national television interview. All questionnaires will be administered via the internet. The 21-item BDI-II will be used as the main outcome measure. Secondary outcome measures will include the Brief Symptom Inventory (53-item BSI), the Inventory of Interpersonal Problems (64-item IIP), and the WHOQOL-BREF.

ELIGIBILITY:
Inclusion Criteria:

* access to the internet
* informed consent to participate
* BDI-II score > 13
* if prescribed, constant dosage of medication (depression/anxiety) for 1 month prior and during study

Exclusion Criteria:

* suicide item of BDI ≥ 2
* other psychological treatment during this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2010-12-31 (Actual); Study Completion 2010-12-31 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory - II (BDI-II) | 10 weeks
  Self-report questionnaire, depression symptom severity, scores can range from 0 to 63, with higher scores indicating more severe depression.

SECONDARY OUTCOMES:
Brief Symptom Inventory (53-item BSI) | 10 weeks
  Psychopathology severity self-report measure; minimum value = 0, maximum value = 4 (higher scores indicate more severe psychopathology).
Inventory of Interpersonal Problems (IIP) | 10 weeks
  Self-report measure of interpersonal problems; total score computed as the mean across all items; minimum value = 0, maximum value = 4 (higher scores indicate more severe psychopathology)
WHOQOL-BREF | 10 weeks
  Self-report quality of life measure; scores can range from 0 to 100, with higher scores indicating better quality of life.

OTHER OUTCOMES:
CSQ-8 (Client Satisfaction Questionnaire) | 10 weeks
  Self-report measure of global client satisfaction; scores can range from 1 to 4, with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Berger, Ph.D., Principal Investigator — University of Bern

IPD SHARING:
Plan to Share IPD: No
Contact the PI for requests to use data.

REFERENCES:
- [Result] Berger T, Hammerli K, Gubser N, Andersson G, Caspar F. Internet-based treatment of depression: a randomized controlled trial comparing guided with unguided self-help. Cogn Behav Ther. 2011;40(4):251-66. doi: 10.1080/16506073.2011.616531. PMID 22060248